CLINICAL TRIAL: NCT06468904
Title: Efficacy of Cervical Stabilization Exercises on Hand Grip Strength, Pinch Strength, Pain Pressure Threshold in Patients With Chronic Myofascial Neck Pain
Brief Title: Efficacy of Cervical Stabilization Exercises on Hand Grip Strength in Chronic Myofascial Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Alzahraa Mohamed Ali Ramadan, principle invesyigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004710
Record Dates: First submitted 2024-06-05; First posted 2024-06-21 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Chronic Neck Pain
Keywords: cervical stabilization; hand grip; myofascial neck pain

STUDY DESIGN:
Intervention Model Description: cervical stabilization exercises
Who Masked: Investigator, Outcomes Assessor
Masking Description: double (investigator, outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical stabilization exercises and integrated neuromuscular inhibition technique (Experimental): patients received cervical stabilization exercises and integrated neuromuscular inhibition technique for 3 sessions / week for 4 weeks. Cervical stabilization included chin tucks, isometric holds, ball squeeze.
  Integrated neuromuscular inhibition technique included:
  1. ischemic compression: therapist applied an intermittent ischemic compression on upper trapezius trigger point by thumb for 90sec.
  2. Strain counter-strain: therapist applied pressure at trigger point. patient's head was laterally flexed towards the affected side passively by one hand of the therapist. The other hand held the subject's forearm and moved the affected shoulder to 90degree of abduction and external rotation for 90 secs.
  3. Muscle energy technique: patient laterally flexed the neck to opposite side patient was moved the stabilized shoulder and ear towards each other. The contraction was maintained for 10 sec followed by 5 seconds of relaxation. The muscle was stretched for 30 secs.
  Interventions: Procedure: cervical stabilization exercises and integrated neuromuscular technique.
- Integrated neuromuscular inhibition technique (Active Comparator): patients received integrated neuromuscular inhibition technique for 3 sessions / week for 4 weeks.it included Ischemic compression, Strain counter-strain and muscle energy technique.
  1. ischemic compression. therapist applied an intermittent ischemic compression on upper trapezius trigger point by thumb for 90 sec.
  2. Strain counter-strain: therapist applied pressure at trigger point. patient laterally flexed towards the affected side passively by one hand of the therapist. The other hand held the subject's forearm and moved the affected side shoulder passively to 90degree of abduction and external rotation for 90 secs.
  3. Muscle energy technique: patient was asked to laterally flex the neck to opposite side. patient was requested to move the stabilized shoulder and ear towards each other. The contraction was maintained for 10 sec followed by 5 seconds of relaxation. The muscle was stretched for 30 secs.
  Interventions: Procedure: cervical stabilization exercises and integrated neuromuscular technique.

INTERVENTIONS:
Procedure: cervical stabilization exercises and integrated neuromuscular technique. — Patients received cervical stabilization exercises and integrated neuromuscular inhibition technique. Cervical stabilization protocol included strengthening exercises of deep cervical flexors muscles which included chin tucks, isometric holds, ball squeeze, as well as deep cervical extensors muscles which included cranio-cervical flexion from neutral, upper cervical rotation and extension of cervical spine.
  integrated technique includes ischemic compression, muscle energy technique and strain counter strain.

SUMMARY:
The purpose of this study is to examine effect of cervical stabilization exercises on hand grip strength, key pinch strength, pain intensity, pain pressure threshold and hand function in chronic myofascial neck pain patients.

DETAILED DESCRIPTION:
Myofascial pain of the trapezius is considered one of the main causes of neck pain and characterized by deep, intense pain of the skeletal muscles and their fascia and by the presence of one or more MTrPs, Although MTrPs can be formed in any muscle or muscle group, previous studies concluded that the upper trapezius(UT) muscle is the most commonly affected muscle.

Considering the role of synergistic function of the UT muscle in scapula-humeral rhythm during shoulder movement, it is not surprising that MTrPs in UT muscle can result in shoulder dysfunction and disability. Muscle activity of proximal parts is necessary for activation of distal parts. In fact, the stable activity of distal parts needs controlling the proximal parts. Thus, the stability of shoulder girdle is required for activity of distal parts such as fingers, wrists and elbows. In addition, trigger points in the UT can affect grip strength, which depends on shoulder joint and scapular stability. Thus, UT muscle dysfunction can reduce grip strength.

However, little research has been carried out to determine the therapeutic effects of cervical stabilization exercises on chronic neck pain, and up till now, there is a gap in literature to explore efficacy of cervical stabilization exercises on chronic neck pain and hand grip strength. Therefore, this study aims to investigate whether cervical stabilization exercises has an effect on hand grip strength in chronic myofascial neck pain.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic neck pain for more than 3 months.
2. Active MTrPs in the UT muscle with a tender nodule.
3. Constant neck pain, a jump sign during palpation of UT muscle.
4. Referred pain.
5. Symptoms of ipsilateral hand muscles weakness.

Exclusion Criteria:

1. Signs of severe pathology such as malignancy of the cervical area.
2. Fractures of the cervical spine.
3. Cervical radiculopathy or myelopathy.
4. Diabetes.
5. Trauma, congenital anomalies and surgery around neck, shoulder and hand.
6. Fibromyalgia or vascular syndromes such as vertebra-basilar insufficiency.
7. Pregnancy.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
primary outcome measure | up to four weeks
  hand grip strength was measured by hand held dynamometer.

SECONDARY OUTCOMES:
secondary outcome measures | up to four weeks
  pain pressure threshold was measured by pressure algometer.
secondary outcome measure | up to four weeks
  hand function was measured by michigan quesstionaire.The Michigan Hand Outcomes Measure comprises 37 items with rating scale ranging 1 to 5. Every single domain was scored and converted to values that range from 0-100. A high score indicates better results, with the exception of pain in which a high score indicates a more intense pain.
secondary outcome measure | up to 4 weeks
  pain intensity was measured by visual analogue scale.The level of pain on the VAS was recorded on a 10 cm line distinct at one end 'no pain' and marked at the other end 'the worst pain. Subjects were asked to state their pain level by placing a mark on this horizontal line
secondary outcome measure | up to four weeks
  pinch strength was measured by pinch gauge

CONTACTS AND LOCATIONS:
Overall Officials: soheir sh Rezkallah, PHD, Study Director — professor of physaical therapy; Ghada Abd Elmoneim, PHD, Study Director — assistant professor of physical therapy; Haidy S Roshdy, PHD, Study Director — lecturer of physical therapy
Locations (2):
- Egypt (2):
  - Cairo University, Giza
  - Faculty of physical therapy, Giza

IPD SHARING:
Plan to Share IPD: No